CLINICAL TRIAL: NCT06168890
Title: Predictive Role of [11C] Choline PET/CT on Survival in Prostate Cancer Patients With Biochemical Failure.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: PETCT-CHOL
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET/CT with choline in the restaging phase of prostate cancer. — PET/CT with choline in the restaging phase of prostate cancer in patients suffering from prostate cancer with biochemical recovery of the disease during hormonal therapy.

SUMMARY:
Several studies have shown that the PET/CT study with Choline is of great use in the restaging of patients with prostate cancer who present a recurrence of biochemical disease following primary treatment. Despite the large amount of literature in which the diagnostic accuracy of the method is highlighted in the identification of the recurrence of prostatic disease both in the case of local recurrence, lymph node recurrence and metastatic disease, there are to date no studies that evaluate whether PET /CT with choline may predict survival in patients radically treated for prostate cancer. The aim of the study is to evaluate the predictive role of choline PET/CT on the survival of patients with biochemical recovery of the disease during hormonal therapy.

This retrospective study will include adult patients affected by prostate cancer with biochemical recurrence of the disease following radical prostatectomy treatment and undergoing hormonal therapy who underwent, between 2004 and 2007, a PET/CT study with choline for the restaging of their disease.

The expected result is to establish how PET/CT with Choline can predict survival in patients who develop a biochemical recurrence of the disease during hormonal therapy. If this result is confirmed, PET/CT with Choline could be even more useful in the follow-up of patients radically treated for prostate cancer to plan the best therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been treated with radical prostatectomy;
* patients who present a progressive increase in PSA value during hormonal treatment.

Exclusion Criteria:

* patients< 18 years

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering from prostate cancer with biochemical recovery of the disease during hormonal therapy who have undergone PET/CT with choline for restaging of the disease after primary treatment.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2014-02-25 (Actual); Study Completion 2014-02-25 (Actual)

PRIMARY OUTCOMES:
PET CT with choline on the survival of patients with biochemical recovery of prostate cancer | 1 year
  PET CT with choline on the survival of patients with biochemical recovery of the disease during hormonal therapy.

IPD SHARING:
Plan to Share IPD: No